CLINICAL TRIAL: NCT05202496
Title: Effect of Oral Systemic Administration of Vitamin D on the Rate of Orthodontic Tooth Movement - A Randomized Control Trial
Brief Title: Effect of Systemic Administration of Vitamin D on the Rate of Orthodontic Tooth Movement - A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dr Revathi M N
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Angle Class I
MeSH Terms: conditions — Malocclusion, Angle Class I | interventions — Calcitriol; Capsules; Orthodontics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: oral vitamin D supplementation during orthodontic treatment (Experimental): The biological methods include using various chemicals like parathyroid hormone, thyroid hormone, prostaglandins, corticosteroids, relaxin and vitamin D.
  Due to its important role in bone remodeling, vitamin D is hypothesized to play an important role in accelerating orthodontic tooth movement.
  experimental group subjects with serum vitamin D levels in the range of 30-40 ng/ml are enrolled
  Interventions: Drug: Calcitriol 0.25Mcg Cap; Procedure: orthodontic treatment
- control : Orthodontic treatment with no intervention (Active Comparator): control group subjects with serum vitamin D levels in the range of (30-40 ng/ml) are enrolled
  Interventions: Procedure: orthodontic treatment

INTERVENTIONS:
Drug: Calcitriol 0.25Mcg Cap — After orthodontic levelling and alignment, experimental group subjects are administered one capsule of calcitriol 0.25 mcg on a daily basis during the study period. Also, serum vitamin D levels are monitored at monthly intervals and rate of canine retraction is measured at monthly intervals
  Other Names: Rocaltrol
  Arms: Experimental: oral vitamin D supplementation during orthodontic treatment
Procedure: orthodontic treatment — experimental group subjects undergo orthodontic treatment after extraction of premolars

SUMMARY:
This study is to evaluate the effect of vitamin D on the rate of tooth movement by measuring and comparing the extraction space closure during retraction in experimental (vitamin D supplemented) and control groups with a sample size of 24 and having serum vitamin D level (30-40 ng/ml). All subjects undergo orthodontic levelling and alignment after premolar extractions followed by vitamin D supplementation in the experimental group. The rate of canine retraction will be measured in both the groups and CBCT taken in the interval of 6 months before and after intervention to measure root changes

DETAILED DESCRIPTION:
Aims and Objectives: To evaluate the effect of vitamin D on the rate of tooth movement by measuring and comparing the extraction space closure during retraction in experimental (vitamin D supplemented) and control groups. Secondary objective: To compare root resorption in experimental and control group. Setting: Department of Orthodontics and Dentofacial Orthopaedics, PGIDS, Rohtak.

Study Design: Prospective, double blind, randomized clinical study Time frame: Duration of study is one year Population/participant: Inclusion criteria:- Patients with age between 19-25 years with malocclusion requiring bilateral extraction of maxillary 1st premolars in good general health and healthy periodontium.

Exclusion Criteria:- Presence of any systemic/bone/metabolic/hormonal diseases, long-term drug history, pregnant or lactating women, smoking habit, root resorption orany chronic disorders Sample size: A sample size of 10 per group for the present study was calculated to detect a clinical difference of 0.89 with a pooled standard deviation of 0.53 (effect size 1.67) at 95% power and alpha significance level at 0.05.

To compensate for 20% dropouts the final sample size was calculated to be 11 per group (i.e) total sample size will be 24.

Method of study: Patients who fulfill the selection criteria will be selected for the study. After taking the pretreatment records and recording the pretreatment vitamin D levels the patients will be sent for extraction of 1st premolars. Treatment will be initiated by bonding 0.022"slot MBT straight wire appliance. Retraction will be done on 0.019"x 0.025" SS wires using closed coil NiTi springs. Patients of study group will be instructed to take adequate dose of vitamin D3 during phase of space closure. Serum vitamin D levels will be checked at 4th,8th, 12th and 16th weeks and rate of canine retraction will be measured at these time intervals. Root resorption will be measured from CBCT at the end of 6 months Outcome Measures: The outcome variables will be the rate of retraction measured in millimeters. Changes in root length will be measured and compared between the two groups Statistical Analysis: Data will be checked for normality. If it is in normal distribution, intra group comparison will be done by student's t-test between two time points and inter group comparison will be done by using Independent T test between two groups. If it is in non-normal distribution, intra group comparison will be done by Wilcoxon signed rank test and inter group comparison will be done by Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

1. Patient in the age group of 19-25 years .
2. Good general health status.
3. Healthy periodontium
4. Absence of root resorption.
5. Absence of any chronic disorders
6. No history of orthodontic treatment.

Exclusion Criteria:

1. Presence of any signs and symptoms of gingival and periodontal diseases.
2. Any Systemic/Bone/metabolic/hormonal disease illness known to affect the outcome of orthodontic therapy or requiring administration of vitamin D
3. Any kind of prolonged drug administration (chronic drug intake)
4. Pregnant or lactating women.
5. Smoking habit.

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Measurement of rate of canine retraction | 4th week
  Distal movement of maxillary canine is measured in mm with the help of electric digital caliper after beginning of maxillary canine retraction
Measurement of rate of canine retraction | 8th week
  Distal movement of maxillary canine is measured in mm with the help of electric digital caliper after beginning of maxillary canine retraction
Measurement of rate of canine retraction | 12th week
  Distal movement of maxillary canine is measured in mm with the help of electric digital caliper after beginning of maxillary canine retraction
Measurement of rate of canine retraction | 16th week
  Distal movement of maxillary canine is measured in mm with the help of electric digital caliper after beginning of maxillary canine retraction

SECONDARY OUTCOMES:
Measurement of Root resorption | 6 months
  Root resorption is measured in relation to canine with the help of CBCT taken before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Sharma, MDS, Study Chair — PGIDS,ROHTAK
Locations (1):
- Pgids,Rohtak, Rohtak, Haryana, India